CLINICAL TRIAL: NCT00003158
Title: A Phase II Trial of Concurrent Carboplatin/VP-16 and Radiation Followed by Paclitaxel (Taxol) for Poor-Risk Stage III Non-Small Cell Lung Cancer
Brief Title: S9712: Radiation Therapy and Combination Chemotherapy in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065951; S9712 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Etoposide; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: etoposide
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy and chemotherapy consisting of carboplatin, etoposide and paclitaxel in treating patients with newly diagnosed stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the survival and failure-free survival in poor risk patients with stage IIIA or IIIB non-small cell lung carcinoma treated with concurrent radiation, carboplatin, and etoposide followed by consolidation with paclitaxel. II. Evaluate the response and toxicities associated with this regimen in this group of poor risk patients.

OUTLINE: This is nonrandomized study. Chemotherapy on cycle 1 starts on day 1 with concurrent initiation of radiotherapy. Chemotherapy is given prior to radiotherapy on those days when both treatments are given. Cycle 2 begins on day 29. Carboplatin is administered by 15 minute IV infusions on days 1, 3, 29, and 31. Etoposide (VP-16) is administered after carboplatin by 30 minute IV infusions on days 1-4, and 29-32. Radiation therapy begins within 24 hours of day 1, cycle 1 of chemotherapy. The primary tumor, the adjacent mediastinum, and other targeted lymph nodes are administered radiotherapy daily 5 days a week for 6.5 weeks. After the 2 cycles of chemotherapy and chest radiotherapy, patients who have stable disease, partial response, or complete response receive 3 cycles of paclitaxel. Paclitaxel is administered by 3 hour IV infusions starting 4 weeks after completion of chemotherapy and radiotherapy and repeated every 3-4 weeks (approximately days 71, 92, and 103) for a total of 3 cycles. Patients are followed every month for the first year, every 3 months for the second year, every 6 months for the third year, and then annually thereafter while on treatment. After treatment, patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: There will be 80 patients accrued in this study over 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed newly diagnosed single primary bronchogenic non-small cell lung cancer (NSCLC) Stage IIIA (T1-2 N2 M0; T3 N0-2 M0) or IIIB (T4 or N3 M0, excluding malignant pleural effusion) Following NSCLC cellular types are eligible: adenocarcinoma large cell carcinoma squamous cell carcinoma unspecified Histology or cytology from involved mediastinal or supraclavicular nodes are sufficient for diagnosis if a separate primary lesion of the lung parenchyma is clearly evident on radiographs Radiographic evidence of mediastinal lymph nodes of at least 1.5 cm in the largest diameter is sufficient to stage N2 or N3 If the largest mediastinal nodes are less than 1.5 cm in diameter and this is the basis for stage III disease, then at least one of the nodes has to be proven positive cytologically or histologically No bronchioloalveolar carcinoma or stage IIIB tumor involving the superior sulcus Patients must meet at least one of the following conditions: - FEV1 less than 2 liters and predicted FEV1 of the contralateral lung no greater than 800 mL based on the quantitative split function testing - Creatinine clearance less than 50 mL/min - Significant clinical hearing loss and unwilling to accept the potential for worsening due to cisplatin - Controlled congestive heart failure that, in the opinion of the investigator, may become decompensated due to excessive hydration prior to cisplatin administration - SWOG performance status 2 and either albumin less than 0.85 times upper limit of normal or weight loss of greater than 10% due to tumor Measurable or evaluable disease Patients with pleural effusion are eligible only if: - pleural fluid must be a transudate with negative cytology if present before mediastinoscopy or exploratory thoracotomy - pleural fluid can be either transudate or exudate with negative cytology if present only after exploratory or staging thoracotomy but not before - in any case, pleural effusion is present only on CT scan but not on decubitus chest x-ray, and it is deemed too small to tap under either CT or ultrasound guidance

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,200/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal SGOT no greater than 1.5 times upper limit of normal Renal: Creatinine clearance at least 20 mL/min Cardiovascular: No unstable congestive heart failure No active angina No unstable cardiac arrhythmias Pulmonary: FEV1 at least 1.0 liter Also See Disease Characteristics Other: No uncontrolled peptic ulcer disease No active infection No prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for 5 years Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiation for lung cancer Surgery: No prior surgery for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 1998-02; Primary Completion 2002-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derick H. Lau, MD, Study Chair — University of California, Davis
Locations (86):
- United States (86):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Davies AM, Chansky K, Lau DH, Leigh BR, Gaspar LE, Weiss GR, Wozniak AJ, Crowley JJ, Gandara DR; SWOG S9712. Phase II study of consolidation paclitaxel after concurrent chemoradiation in poor-risk stage III non-small-cell lung cancer: SWOG S9712. J Clin Oncol. 2006 Nov 20;24(33):5242-6. doi: 10.1200/JCO.2006.07.0268. PMID 17114656
- [Result] Davies AM, Lau DH, Crowley J, et al.: Concurrent carboplatin/etoposide and radiation followed by paclitaxel consolidation for poor risk stage III non-small cell lung cancer: a Southwest Oncology Group (SWOG) phase II trial (S9712). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1191, 2002.